CLINICAL TRIAL: NCT01756170
Title: Phase III Randomized Trial of Comparing Chemoradiotherapy vs. Radiotherapy Alone in Lymph Node Negative Patients With Early-Stage Cervical Cancer Following Radical Hysterectomy
Brief Title: Postoperative Chemoradiation v.s Radiotherapy for Lymph Node Negative Cervical Cancer Patients
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: xie congying (Other)
Responsible Party: Sponsor-Investigator, xie congying, Director, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WZMC-11352
Record Dates: First submitted 2012-12-13; First posted 2012-12-25 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Cervical Cancer
Keywords: cervical cancer; radiotherapy; postoperative therapy; chemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Paclitaxel; Cisplatin; Radiotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 2 (Active Comparator): Patients receive radiotherapy alone as in arm 1.
  Interventions: Radiation: Radiotherapy
- Arm 1 (Experimental): Patients in this arm will postoperatively receive paclitaxel 135 mg/m2 d1 and cisplatin 25mg/m2 d1-3 intravenously every 4 weeks with radiation. Radiotherapy consisted of 46-50 gray (5 x 2.0 gray/week) on pelvic area.
  Interventions: Drug: paclitaxel; Drug: cisplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: paclitaxel
  Arms: Arm 1
Drug: cisplatin
  Arms: Arm 1
Radiation: Radiotherapy

SUMMARY:
This phase III study is designed to examine if low-risk (lymph node negative), stage I a2-II b cervical cancer patients treated by paclitaxel/cisplatin chemoradiation have greater toxicities but similar survival rate as those treated by radiotherapy alone.

DETAILED DESCRIPTION:
Cervical carcinoma is one of the most common gynecologic cancers worldwide. Concurrent radiotherapy with cisplatin-based chemotherapy has become the standard treatment for patients with high risk factors cervical cancer. However, the treatment modality in patients with low-risk (lymph node negative) is still disputable. It is not yet known whether cisplatin-based chemoradiotherapy are more effective than radiotherapy alone in treating these patients.

Therefore, the investigators are going to perform the efficacy and safety study of postoperative concurrent paclitaxel/cisplatin chemoradiotherapy vs. radiotherapy alone in lymph node negative patients with early-stage cervical cancer following radical hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Undertaken radical hysterectomy with diagnosis of invasive cervical cancer (non-small cell type)
* Negative lymph node
* At least two risk factors (interstitial infiltration of greater than 1/3, vascular or lymphatic involvement, cervix neoplasms larger than 4 cm, nerve involvement)
* Eastern Cooperative Oncology Group 0-2
* Expected life span over 6 months.
* No distant metastasis
* Adequate bone marrow functions (absolute neutrophil count≥ 1,500/ul, blood platelet≥ 100,000/ul, haemoglobin≥ 10g/dl)
* Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
* Adequate liver functions (serum bilirubin ≤ 1.5mg/dl, aspartate aminotransferase/alanine aminotransferase ≤ 3 times(normal value)
* Written informed consent

Exclusion Criteria:

* Previous history of chemotherapy or radiation
* Hypersensitive reaction to platinum/paclitaxel agent
* History of other cancer
* Concurrent systemic illness not appropriate for chemotherapy
* Active infection requiring antibiotics
* Pregnancy

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
disease-free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 5 years

OTHER OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 1 year
  assessed by NCI Common Terminology Criteria v3.0

CONTACTS AND LOCATIONS:
Overall Officials: Congying Xie, MD, Study Director — the 1st Affiliated Hospital of Wenzhou Medical College
Locations (1):
- The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China